CLINICAL TRIAL: NCT05548660
Title: Pharmacogenetic-guided Choice of Post-surgery Analgesics
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sony Tuteja, Research Assistant Professor of Medicine, Division of Translational Medicine and Human Genetics; Assistant Director, Pharmacogenomics Penn Center for Precision Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 851447
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Pain; Post Operative Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Post-surgery pharmacogenetic-guided analgesic selection versus usual care analgesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGx-guided (Experimental): Pharmacogenetic testing using a 16 gene panel with a pharmacist consult providing genotype-guided recommendations for post-surgery analgesic selection based on CYP2D6 and CYP2C9 results. Pharmacist recommendations for all 16 gene results will also be provided in a detailed note.
  Interventions: Other: Pharmacogenetic testing; Other: Pharmacist note with genotype-guided analgesic recommendations; Other: Pharmacist detailed note with genotype-guided recommendations per CPIC guidelines
- Usual care (Other): Pharmacogenetic testing using a 16 gene panel. Post-surgery analgesic selection will be based on usual care (not the PGx results). Pharmacist recommendations for all 16 gene results will be provided in a detailed note with a delayed return of results (30 days post surgery)
  Interventions: Other: Pharmacogenetic testing; Other: Pharmacist detailed note with genotype-guided recommendations per CPIC guidelines

INTERVENTIONS:
Other: Pharmacogenetic testing — Genetic testing of CYP2B6, CYP2C19, CYP2C9, CYP2C cluster CYP2D6, CYP3A5, CYP4F2, DPYD, HLA-A, HLA-B, IFNL4, NUDT15, SLCO1B1, TPMT, UGT1A1, and VKORC1.
Other: Pharmacist note with genotype-guided analgesic recommendations — CYP2C9 normal metabolizers will be recommended to receive ibuprofen and intermediate and poor metabolizers will be recommended to receive naproxen.
  CYP2D6 normal metabolizers will be recommended to receive tramadol and ultrarapid, intermediate and poor metabolizers will be recommended to receive oxycodone.
  Arms: PGx-guided
Other: Pharmacist detailed note with genotype-guided recommendations per CPIC guidelines — Genotype-guided recommendations for all actionable phenotypes resulted from the 16-gene PGx panel per CPIC guidelines and FDA labeling

SUMMARY:
Pharmacogenomics (PGx) is the study of how genes affect a person's response to drugs. PGx testing for certain genes can help predict the risk of side effects or therapeutic failure from analgesics. Testing is not regularly performed in clinical practice due to long wait times for results and challenges with integrating test results in the electronic health record. Investigators leading this study hope to find out if providing surgeons with the ability to order a PGx test and electronically receive results with dosing recommendations will increase the use of these tests to guide analgesic choice and improve patient outcomes.

This is a prospective, two-arm randomized implementation study. Eligible participants will be randomly assigned to receive genotype-guided analgesic selection (intervention arm) or usual care (control arm). Both cohorts will undergo pharmacogenetic testing at the time of consenting. The investigators will primarily measure the feasibility of using this test to guide analgesic selection.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent
2. Assigned female at birth and aged 18 years or older at the time of study initiation
3. Major gynecologic surgery indicated and planned for hysterectomy, myomectomy, exploratory laparotomy, and open abdominal surgery
4. Willing to provide a buccal swab for PGx testing and comply with all study-related procedures

Exclusion Criteria:

1. Receiving chronic opioid therapy defined as ≥ 3 consecutive months of 1-month prescriptions for an opioid
2. Pregnancy
3. Breastfeeding
4. Treating physician does not want subject to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of integrating a PGx panel test in the EMR with a pharmacist consult note for each patient | 14 days
  The proportion of PGx test results and pharmacist consult notes returned prior to surgery
Fidelity to genotype-guided pharmacotherapy recommendations | 14 days
  The proportion of medication selections made in agreement with the genotype-guided dosing recommendations for analgesic medications.

SECONDARY OUTCOMES:
Acute pain - Self-reported numeric pain score | 14 days
  Mean patient self-reported numeric pain scores (scale: 0-10, 0 = no pain; 10= worst pain imaginable) assessed on POD 0, 3, 7, 14 in the PGx-guided group vs. the control group
Total opioid consumption in morphine milligram equivalents (MME) | 14 days
  Difference in total MME consumption in variant carriers in PGx-guided group vs. control group

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, ICF will be made available 1 year following enrollment of the last participant. IPD will be made available 6 months after publication of study results
Access Criteria: Contact PI, Sony Tuteja, PharmD, sonyt@pennmedicine.upenn.edu with individual requests.